CLINICAL TRIAL: NCT05695820
Title: Effects of Low- Load Strengthening Using Different Exercises Modes During Blood Flow Restriction for Treating Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Gad Moussa, Msc degree in physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004174
Record Dates: First submitted 2023-01-11; First posted 2023-01-25 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Blood flow restriction/ shoulder impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Parallel Groups Clinical Trial
Who Masked: Participant
Masking Description: Sealed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Concentric (Experimental): Concentric group
  Interventions: Other: Blood Flow Restriction training
- Isometric (Experimental): Isometric group
  Interventions: Other: Blood Flow Restriction training
- Eccentric (Experimental): Eccentric group
  Interventions: Other: Blood Flow Restriction training

INTERVENTIONS:
Other: Blood Flow Restriction training — It is a method that involves reducing blood flow to a muscle by the application of an external constricting device, such as a blood pressure cuff or tourniquet, to provide mechanical compression of the underlying blood vessels. BFR is applied aiming to enhance blood pooling in the capillary beds of the limb muscles distal to the tourniquet

SUMMARY:
Purpose of the study: This study compares effects of isometric, concentric and eccentric exercises for shoulder muscles by using low load blood flow restriction training on pain, strength and function in patients with SIS.

DETAILED DESCRIPTION:
This study will be conducted at El hadra university hospital, Alexandria, Egypt. Study Design: Randomized Parallel Groups Clinical Trial. Participants: Sixty patients of both genders with unilateral shoulder impingement syndrome, with age range from 30-40 years will be randomly assigned to 1 of 3 groups. All patients will be referred by the orthopedic surgeon who will diagnose shoulder impingement syndrome based on clinical and radiological examination. Group 1: twenty patients will receive concentric training of rotator cuff muscles while applying blood flow restriction for 4 weeks. Group 2: twenty patients will receive eccentric training of rotator cuff muscles while applying blood flow restriction for 4 weeks. Group 3: twenty patients will receive isometric training of rotator cuff muscles while applying blood flow restriction for 4 weeks. The assessment for all groups will be done at baseline and after 4 weeks.

ELIGIBILITY:
Inclusion criteria:

Age range 30-40 years. - Pain localized to the proximal anterolateral shoulder region, - Positive for pain on at least one of the following three impingement tests: Hawkins-Kennedy, Neers, Jobes and Positive for pain on at least one of the following four tests: Painful arc, drop arm test, lift off test, and resisted external rotation (Fatima et al., 2021

Exclusion Criteria:

* Large, full-thickness rotator cuff tear, Moderate, severe glenohumeral or acromioclavicular joint osteoarthritis. - Glenohumeral joint instability including previous shoulder dislocation/subluxation. - Previous shoulder fracture. - Current neck pain/dysfunction with a somatic or radicular referral pattern indicative of cervical spine rather than shoulder as primary source of symptoms and/or pathology. - Neurological deficits of the upper limb. - Systemic inflammatory arthritic conditions (Fatima et al., 2021).

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 20 minutes
  All HHD assessments will be done in the form of three trials of 3 seconds of maximal isometric contraction and a 10-second rest period between each measurement. The mean peak force, will be recorded in kilograms (Kgs), and used as the strength measure

SECONDARY OUTCOMES:
Functional assessment | 20 minutes
  By DASH questionnaire
Pain assessment | 15 minutes
  By visual analogue scale
Range of motion | 20 minutes
  By bubble inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ma Gad, Study Director — Cairo University
Locations (1):
- CairoU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Website